CLINICAL TRIAL: NCT06940726
Title: Exploration Des Liens Entre Audition, Cognition et activité cérébrale Chez Des Personnes présentant un acouphène
Brief Title: Exploring the Links Between Hearing, Cognition and Brain Activity in People With Tinnitus
Acronym: GHOSTTONE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: IHU reConnect (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-159; 2025-A00267-42 (Other: ID-RCB)
Record Dates: First submitted 2025-04-08; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-03

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Hearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Sham Comparator)
  Interventions: Other: Quality of Life questionnaires; Other: Hearing tests; Behavioral: Auditory prediction task; Behavioral: Attention task
- Subjets with tinnitus (Experimental)
  Interventions: Other: Quality of Life questionnaires; Other: Hearing tests; Behavioral: Auditory prediction task; Behavioral: Attention task

INTERVENTIONS:
Other: Quality of Life questionnaires — Subjects will complete a number of self-questionnaires on subjects such as attention span, anxiety levels and sleep quality.
Other: Hearing tests — listening to sounds on headphones and repeating words
Behavioral: Auditory prediction task — listening to sounds and assessing auditory perception
Behavioral: Attention task — assessment of reaction time to visual or auditory cues

SUMMARY:
The goal of this observational study is to understand the mechanisms underlying tinnitus, and improve the clinical assessment strategies needed to develop targeted therapeutic interventions by comparing endogenous attention capacities in healthy subjects and subjects with tinnitus

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Good written and oral comprehension of the French language
* Normal or corrected vision

Group of people with tinnitus :

- Chronic tinnitus > 3 months, uni or bilateral, stable (no period of remission)

Control group :

- No tinnitus

Exclusion Criteria:

* Presence of a known neurological disorder
* Presence of a known degenerative pathology
* Presence of a known hearing impairment
* Presence of a motor disability of the upper limbs
* Severe or profound deafness on one or both sides
* Person under legal protection (guardianship, curatorship, etc.)
* Use of hearing aids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Contingent negative variation (CNV) in EEG | 2 hours

SECONDARY OUTCOMES:
Response reaction time (in ms) | 2 hours
  Comparison of reaction time (RT) variability following response button presses in behavioural tasks
Answer accuracy (% correct answers) | 2 hours
  Comparison of the variability of the number of correct responses following button presses in behavioural tasks.
Cerebral oscillations (alpha bands) obtained by EEG during behavioural tasks | 2 hours
Skin conductance (μS) | 2 hours
  during behavioral task
Heart rate variability (in ms) | 2 hours
  during behavioral task
Pupillometry (pupillary dilation in mm) | 2 hours

IPD SHARING:
Plan to Share IPD: Undecided